CLINICAL TRIAL: NCT02391142
Title: Clinical Assessment of the Treatment With Cardiac Sympathetic Blockade on Chronic Heart Failure
Acronym: CSB-CHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSB-CHF
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2014-05

CONDITIONS: Heart Failure
Keywords: heart failure; cardiac sympathetic nerve block; sympathetic nervous system
MeSH Terms: conditions — Heart Failure | interventions — Lidocaine; Ropivacaine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- cardiac sympathetic nerve block (Experimental): lidocaine or ropivacaine epidural injection
  Interventions: Drug: Lidocaine
- non-cardiac sympathetic nerve block (No Intervention)

INTERVENTIONS:
Drug: Lidocaine — 0.5% lidocaine 5ml epidural injection every 2 hours per day or 0.2% ropivacaine 5ml epidural injection every 4 hours per day, last for 4weeks
  Other Names: ropivacaine
  Arms: cardiac sympathetic nerve block

SUMMARY:
The purpose of this study is to evaluate the effect of Cardiac Sympathetic Blockade on Mortality, re-hospitalization rate, symptoms, quality of life, exercise tolerance, cardiac structure, systolic function, electrical activities and concentration of B - type natriuretic peptide precursor in patients with Chronic Heart Failure.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years old
* more than 3 months of chronic heart failure history or clinical symptoms of heart failure last for more than 3 months (including acute episode of chronic heart failure), chronic heart failure diagnostic criteria refer to 2012ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure
* NYHA functional class III-IV, ejection fraction ≤45%
* NT-proBNP>400ng/L

Exclusion Criteria:

* first episode of acute heart failure
* unrepaired valvular heart disease accompanied with Hemodynamic changes
* hypertrophic cardiomyopathy, pericardial disease, congenital heart disease, severe pulmonary hypertension
* Second-degree type 2 or worse sinoatrial or atrioventricular block without pacemaker therapy
* right heart failure caused by various diseases, respiratory failure or right heart failure induced by chronic obstructive pulmonary disease
* overt renal decompensation: serum creatinine>2.1mg/dl(186umol/L)
* severe hepatic dysfunction, transaminase or alkaline phosphatase > 3 times the upper limit of normal
* Cerebral vascular accident in three months( cerebral infarction, cerebral embolism, cerebral hemorrhage,etc)
* life expectancy shorter than 6 months
* patients with a previous or present history of tumour or precancerous lesions confirmed by pathological examination
* Spine Deformity or skin infection at puncture site
* participate in any clinical drug trials in the three months
* the patients who do not sign the informed consent, unable or unwilling to comply with the requirements of the protocol or unsuitable for the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | one year

SECONDARY OUTCOMES:
Rehospitalization rate | one year

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China